CLINICAL TRIAL: NCT01866345
Title: Randomized, Blinded, Controlled Clinical Trial of Surgically Facilitated Orthodontic Treatment in the Mandibular Anterior Region
Brief Title: Randomized, Blinded, Controlled Clinical Trial of Surgically Facilitated Orthodontic Treatment
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Cannot find subjects to particpate
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1305M32543
Record Dates: First submitted 2013-05-28; First posted 2013-05-31 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Orthodontic Malocclusion
Keywords: orthodontics; Tooth Movement; Bone Remodeling; Mandible; Osteotomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional orthodontic treatment (Active Comparator): conventional orthodontic treatment in the mandibular anterior region
  Interventions: Procedure: Conventional orthodontic treatment
- Surgically facilitated Orthodontics (Experimental): Surgically facilitated Orthodontic treatment in the mandibular anterior region
  Interventions: Procedure: Surgically facilitated Orthodontic treatment

INTERVENTIONS:
Procedure: Surgically facilitated Orthodontic treatment — Surgically facilitated Orthodontic treatment in the mandibular anterior region
  Arms: Surgically facilitated Orthodontics
Procedure: Conventional orthodontic treatment — Conventional orthodontic Procedure
  Arms: Conventional orthodontic treatment

SUMMARY:
The purpose of this investigation is intended to evaluate the efficacy of surgically facilitated orthodontic treatment (SFO) in terms of treatment time, incidence of root shortening, and occurrence of mucogingival side effects compared to conventional orthodontic therapy in patients undergoing orthodontic treatment to correct crowding and/or retroclination of their mandibular anterior dentition.

DETAILED DESCRIPTION:
The null-hypothesis for this research project is that there will be no difference in the rate of orthodontic movement among patients requiring proclination or alignment of their mandibular anterior teeth with SFO (TEST group) as compared to conventional orthodontic treatment (CONTROL group). A null-hypothesis is that there will be no difference between both treatment groups in the occurrence of dental (root shortening) or periodontal (mucogingival defects, alveolar bone resorption) complications associated with orthodontic treatment.

ELIGIBILITY:
Inclusion Criteria:

-Adults (18-65 y.o.) who seek orthodontic treatment for proclination and/or de-crowding of mandibular anterior teeth.

Exclusion Criteria:

* Bone-related diseases
* Previous or current use of biphosphate therapy
* Previous mucogingival surgery in the area
* Genetic syndromes, craniofacial anomalies, or cleft lip and/or palate

  - History of previous orthodontic treatment less than 4 years ago
* Smoking >10 cigarettes/day )
* Medical history that contraindicates surgical treatment,
* People who are not cognitively able to give consent,
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Rate of orthodontic tooth movement | 6 months(plus or minus 1 week)
  Difference between the rate of orthodontic tooth movement between the two groups as measured by linear measurements on digitized study casts obtained at 4-week intervals.

SECONDARY OUTCOMES:
Incidence of mucogingival defects | 6 months(plus or minus 2weeks) after initiation of treatment
  Incidence of mucogingival defects as clinically measured by gingival recession (GR), clinical attachment level (CAL), probing depth (PD), width of keratinized tissue (WKT) and biotype), by a calibrated examiner
Incidence and magnitude of apical root resorption | 6(plus or minus 1) months following initiation of treatment
  Incidence and magnitude of apical root resorption will be estimated from pre- and post-treatment cone-beam computed tomograms (CBCTs)

OTHER OUTCOMES:
Thickness and height of the buccal and lingual bony plates | 6(plus or minus 1) months following initiation of treatment
  Thickness and height of the buccal and lingual bony plates will be measured from pre- and post-treatment Cone beam volumetric tomograms

CONTACTS AND LOCATIONS:
Overall Officials: Georgios A Kotsakis, DDS, Principal Investigator — Dental Fellow

REFERENCES:
- [Background] Murphy KG, Wilcko MT, Wilcko WM, Ferguson DJ. Periodontal accelerated osteogenic orthodontics: a description of the surgical technique. J Oral Maxillofac Surg. 2009 Oct;67(10):2160-6. doi: 10.1016/j.joms.2009.04.124. No abstract available. PMID 19761909
- [Background] Sebaoun JD, Kantarci A, Turner JW, Carvalho RS, Van Dyke TE, Ferguson DJ. Modeling of trabecular bone and lamina dura following selective alveolar decortication in rats. J Periodontol. 2008 Sep;79(9):1679-88. doi: 10.1902/jop.2008.080024. PMID 18771369